CLINICAL TRIAL: NCT01083368
Title: Phase I-II Study Evaluating the Safety and Clinical Efficacy of Temsirolimus and Avastin in Patients With Chemotherapy Refractory Castrate Resistant Prostate Cancer (CRPC)
Brief Title: Temsirolimus and Bevacizumab in Hormone-Resistant Metastatic Prostate Cancer That Did Not Respond to Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7808; NCI-2010-00308 (Other: NCI/CTRP); CASE7808 (Other: Case Comprehensive Cancer Center); CASE7808-CC527 (Other: Cancer Center IRB)
Record Dates: First submitted 2010-03-05; First posted 2010-03-09 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; hormone-resistant prostate cancer; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — temsirolimus; Sirolimus; Bevacizumab; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: Combination of temsirolimus and AVASTIN (Experimental): Patients receive temsirolimus IV over 30-60 minutes once weekly and bevacizumab IV over 30-90 minutes once every two weeks . Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temsirolimus; Biological: bevacizumab; Genetic: polymorphism analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; rapamycin analog CCI-779; Torisel
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; anti-VEGF rhuMAb; Avastin; recombinant humanized anti-VEGF monoclonal antibody; rhuMAb VEGF
Genetic: polymorphism analysis — Correlative studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving temsirolimus together with bevacizumab may be a better way to block tumor growth.

PURPOSE: This phase I/II trial is studying the side effects and best dose of temsirolimus when given together with bevacizumab and to see how well it works in treating patients with hormone-resistant metastatic prostate cancer that did not respond to chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of the Phase I portion of this study is to determine the maximum tolerated dose (MTD) of temsirolimus in combination with AVASTIN in subjects with chemotherapy refractory metastatic CRPC.

II. The primary objective for the Phase II portion of this study is to evaluate the objective response frequency (PSA and RECIST-Response Evaluation Criteria in Solid Tumors-defined) of the combination of temsirolimus and AVASTIN in patients with chemotherapy refractory metastatic CRPC.

SECONDARY OBJECTIVES:

I. To evaluate the effect of the combination of temsirolimus and AVASTIN on time to clinical progression and overall survival in patients with chemotherapy refractory metastatic CRPC.

II. To further evaluate the safety of temsirolimus given in combination with AVASTIN in chemotherapy refractory metastatic CRPC patients at the dose established in our phase I safety phase.

III. To determine the presence of circulating tumor cells (CTCs) and status of single nucleotide polymorphism (SNPs) in CRPC patients. (Exploratory)

OUTLINE: Patients receive temsirolimus IV over 30-60 minutes once weekly and bevacizumab IV over 30-90 minutes once every two weeks . Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 28 days.

ELIGIBILITY:
Inclusion

* Understand and voluntarily sign an informed consent form
* Patients with histologically confirmed adenocarcinoma of the prostate
* Patients must have evidence of chemotherapy-refractory metastatic CRPC following standard antiandrogen withdrawal (AAWD); CRPC will be defined as patients with metastatic prostate cancer with radiologic evidence of metastases on either bone scan, plain x-rays, CT scans, chest x-ray, and castrate levels of testosterone ( =< 50 mg/dL)
* All patients must be receiving ongoing therapy to ensure testicular androgen suppression (LHRH therapy or bilateral orchiectomy)
* Patients must have received prior Docetaxel-based or Mitoxantrone-based chemotherapy; previous chemotherapy treatments must be completed at least 4 weeks prior to screening, and patients must not have any residual therapy-related toxicity present at screening
* Patients must be off any steroids 7 days prior to the initiation of treatment
* Patients must have evidence of disease progression defined as any of the following:
* a) New sites of metastatic disease on radiographic imaging (bone scan or CT scan of chest/abdomen/pelvis) as determined by the referring physician
* b) PSA progression, defined as 2 consecutive PSA rise at least 2 weeks apart with PSA value over a baseline level of at least 5.0 ng/mL, confirmed after an interval of at least two weeks
* ECOG performance status 0-2 (Eastern Cooperative Oncology Group)
* Absolute neutrophil count >= 1500/uL
* Hemoglobin >= 8 g/dL (blood transfusion not permitted within 2 weeks prior to first dose of treatment)
* Platelets >= 100,000/uL
* Serum creatinine =< 1.5 x ULN
* Total bilirubin =< 1.5 x ULN
* AST (aspartate aminotransferase-SGOT) and ALT (SGPT) that are =< 2.5 x ULN (5 x ULN in patients with liver metastasis)
* Fasting cholesterol =< 350mg/dL and fasting triglycerides =< 400mg/dL
* Hemoglobin A1c (HgbA1c) < 10% (optimal therapy permitted)
* Therapeutic INR/PT for those patients receiving oral anticoagulation
* Urine protein:creatinine ratio (UPC) =< 1.0 at screening
* QTc interval =< 450 msec for males and =< 470 msec for females
* The use of cholesterol medications is allowed during the study
* Patients with a history of a prior malignancy are eligible provided they were treated with curative intent and have been disease-free for the time period considered appropriate by the treating physician
* Sexually active men whose sexual partners are women of childbearing potential must agree to use a medically acceptable form of barrier contraception or abstinence during their participation in the study and for at least six weeks after study drug discontinuation
* Patients on stable doses of bisphosphonates that show subsequent tumor progression may continue on this medication; however, patients are not allowed to initiate bisphosphonate therapy within 4 weeks prior to starting therapy or throughout the study
* Prior radiopharmaceuticals (strontium, samarium) must be completed at least 8 weeks prior to treatment initiation in this study and all major side effects resolved to =< grade 1
* Patients receiving any other hormonal therapy, including any dose of Megestrol acetate (Megace), Proscar (finasteride), any herbal product known to decrease PSA levels (e.g., Saw Palmetto and PC-SPES), must discontinue the agent for at least 4 weeks prior to enrollment
* Life expectancy of at least 12 weeks
* Written informed consent/HIPAA (Health Insurance Portability and Accountability Act)authorization must be provided prior to the performance of any study-related procedures

Exclusion

* Prior treatment with AVASTIN, temsirolimus, everolimus or sirolimus
* Evidence of current or prior central nervous system (CNS) metastases or any imaging abnormality indicative of CNS metastases; patients with history of cord compression are eligible provided they had either palliative radiation therapy or surgery, have NO neurologic symptoms (as determined by treating physician), have stable spinal disease by scans and are off any steroids prior to initiating study drug (at least 7 days)
* Major surgery or radiation therapy within 28 days prior to screening (Palliative radiotherapy to painful bone lesions is allowed within 14 days prior to study entry); subject must have recovered from prior surgery and radiation
* Significant cardiovascular disease defined as congestive heart failure (NYHA Class II, III, or IV), angina pectoris requiring nitrate therapy, or myocardial infarction within the last 6 months
* Inadequately controlled hypertension (defined as a blood pressure of >= 150 mmHg systolic and/or >= 100 mmHg diastolic on medication), or any prior history of hypertensive crisis or hypertensive encephalopathy
* History of stroke or transient ischemic attack within 6 months prior to screening
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection), or symptomatic peripheral vascular disease
* Known congenital long QT syndrome, history of Torsade de pointes or ventricular tachycardia
* Known pulmonary hypertension or pneumonitis
* More than 1 episode of DVT/PE within the last 6 months
* Evidence or history of bleeding diathesis or coagulopathy
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to screening
* Supplements or complementary medicines/botanicals are not permitted while on protocol therapy, except for any combination of the following: conventional multivitamin supplements; selenium; lycopene; soy supplements; patients should review the label with their doctor prior to enrollment, and discontinue disallowed agents prior to study enrollment; patients taking St. John's Wort need to discontinue its use at least 7 days prior to initiating trial
* Serious intercurrent infections or non-malignant medical illnesses including uncontrolled autoimmune disorders
* Psychiatric illnesses/social situations that would limit compliance with protocol requirements
* Known contraindication to receive temsirolimus or AVASTIN
* Use of any other experimental drug or therapy within 28 days of baseline
* Immunocompromised subjects, including known seropositivity for human immunodeficiency virus (HIV), or current or chronic hepatitis B and/or hepatitis C infection (as detected by positive testing for hepatitis B surface antigen [HbsAg] or antibody to hepatitis C virus [anti HCV] with confirmatory testing) (testing is not mandatory to be eligible for the study)
* Anticancer therapies such as biologic therapy and chemotherapy, as well as radiation therapy or cancer surgery
* Other current or recent (within 4 weeks prior to randomization) investigational agent
* Rifampicin
* Immunosuppressive therapies except steroids
* Prophylactic use of white blood growth factors to support neutrophils
* Concomitant treatment with agents that have CYP3A4 induction or inhibition potential should be voided

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Garcia, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Matthew Cooney, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - CCF-Willoughby Hills, Willoughby Hills, Ohio

REFERENCES:
- [Derived] Barata PC, Cooney M, Mendiratta P, Gupta R, Dreicer R, Garcia JA. Phase I/II study evaluating the safety and clinical efficacy of temsirolimus and bevacizumab in patients with chemotherapy refractory metastatic castration-resistant prostate cancer. Invest New Drugs. 2019 Apr;37(2):331-337. doi: 10.1007/s10637-018-0687-5. Epub 2018 Nov 7. PMID 30402678

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from medical clinics from 3/2009 to 7/2011
Pre-assignment Details: 22 participants were enrolled, but only 21 treated because one participant withdrew before start of protocol therapy.
Groups:
- Dose Level -1: Temsirolimus 15 mg IV q wk with Bevacizumab 5 mg/kg IV q 2 wks
  This is a de-escalation dose levels and no participants ended up receiving this dose level.
- Dose Level 0: Temsirolimus 15 mg IV q wk with Bevacizumab 10 mg/kg IV q 2 wks
  This is a de-escalation dose levels, and no participants ended up receiving this dose level.
- Dose Level 1: Temsirolimus 20 mg IV q wk with Bevacizumab 10 mg/kg IV q 2 wks
- Dose Level 2: Temsirolimus 25 mg IV q wk with Bevacizumab 10 mg/kg IV q 2 wks
Period: Dose Escalation Weeks 1-4
Arm/Group | Dose Level -1 | Dose Level 0 | Dose Level 1 | Dose Level 2
Started | 0 | 0 | 4 | 0
Disease Progression | 0 | 0 | 1 | 0
Completed | 0 | 0 | 4 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Dose Escalation Weeks 5-9
Arm/Group | Dose Level -1 | Dose Level 0 | Dose Level 1 | Dose Level 2
Started | 0 | 0 | 1 (Participant on DL1 did not move to dose level 2 because of disease progression.) | 6
Completed | 0 | 0 | 1 | 6 (3 participants on dose level 1 moved to dose level 2, 3 more new participants joined.)
Not Completed | 0 | 0 | 0 | 0
Period: Phase II - Efficacy/Safety
Arm/Group | Dose Level -1 | Dose Level 0 | Dose Level 1 | Dose Level 2
Started | 0 | 0 | 0 | 20
Completed | 0 | 0 | 0 | 20 (14 plus 6 participants from previous period)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only subjects that received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 4 | 17 | 21
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 0 | 5 | 5
  60-69 years | 3 | 5 | 8
  70-79 years | 1 | 6 | 7
  80-89 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 17 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 16 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 4 | 13 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 17 | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Temsirolimus (Phase I)
Description: Participants received temsirolimus (20mg or 25mg IV weekly) in combination with a fixed dose of IV bevacizumab (10mg/kg every 2 weeks). The MTD was determined to be the dose at which no unacceptable toxicities were observed.
Time Frame: at 24 weeks
Population: Subjects that received treatment for the Dose escalation portion of the study.
Measure: Number; unit: mg
Groups:
- Dose Levels 1 and 2: Patients receive temsirolimus IV over 30-60 minutes once weekly and bevacizumab IV over 30-90 minutes once every two weeks . Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  temsirolimus: Given IV
  bevacizumab: Given IV
  polymorphism analysis: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Dose Levels 1 and 2
Number analyzed (Participants) | 6
mg | 25

2. Primary Outcome: Objective Response (Dose Level 2)
Description: PSA (Prostate-Specific Antigen) test will be performed every 4 weeks prior to receiving treatment. PSA response will be measured as the number of participants that had a decline observed from baseline.
Time Frame: change from baseline to 12 weeks
Population: Participants with available serial PSA data (at both baseline and 12 weeks) who received the MTD dose of Temsirolimus 25 mg.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 2: Patients receive temsirolimus IV over 30-60 minutes once weekly and bevacizumab IV over 30-90 minutes once every two weeks . Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Level 2
Number analyzed (Participants) | 16
Participants | 5

3. Secondary Outcome: Time to Clinical Progression
Description: To evaluate the effect of the combination of temsirolimus and AVASTIN on time (in months) to clinical progression from start of treatment. Progressive Disease according to RECIST Criteria is defined as : At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 12 weeks
Population: All participants that received treatment. Data no longer available per intervention arms - reported combined.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Combination of Temsirolimus and AVASTIN: Patients receive temsirolimus IV over 30-60 minutes once weekly and bevacizumab IV over 30-90 minutes once every two weeks . Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  temsirolimus: Given IV
  bevacizumab: Given IV
  polymorphism analysis: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Combination of Temsirolimus and AVASTIN
Number analyzed (Participants) | 21
months | 2.6 [1.2 to 3.9]

4. Secondary Outcome: Overall Survival
Description: Time in months from on study to time of death
Time Frame: baseline to end of study, up to 3.5 years
Population: All participants that received treatment. Data no longer available per intervention arms - reported combined.
Measure: Median (Full Range); unit: months
Arm/Group | Combination of Temsirolimus and AVASTIN
Number analyzed (Participants) | 21
months | 8 [3 to 42]

5. Secondary Outcome: Number of Patients With Toxicity as Assessed by CTCAE v3.0 (Common Toxicity Criteria for Adverse Effects)
Description: To further evaluate the safety of temsirolimus given in combination with AVASTIN in chemotherapy refractory metastatic CRPC patients at the dose established in our phase I safety phase. Specific toxicities are listed in the SAE and AE results.
Time Frame: at 24 weeks
Population: All participants who received treatment at the MTD (Dose level 2)
Measure: Number; unit: participants
Arm/Group | Combination of Temsirolimus and AVASTIN
Number analyzed (Participants) | 17
participants | 17

6. Other Pre Specified Outcome: Presence of Circulating Tumor Cells and Single Nucleotide Polymorphism Status
Description: To determine the presence of circulating tumor cells (CTCs) and status of single nucleotide polymorphism (SNPs) in CRPC patients.
Time Frame: at end of treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Prostate Specific Androgen (PSA)
Description: Prostate Specific Androgen (PSA) at baseline
Time Frame: at baseline
Population: All participants that received treatment for both arms. Data no longer available per intervention arms - reported combined.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Arm 1: Combination of Temsirolimus and AVASTIN
Number analyzed (Participants) | 21
ng/mL | 205.3 [11.1 to 1801.0]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected while participants were on study up to 3 1/2 years.
Groups:
- Dose Level 1: Patients receive temsirolimus IV over 30-60 minutes once weekly and bevacizumab IV over 30-90 minutes once every two weeks . Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  temsirolimus: Given IV
  bevacizumab: Given IV
  polymorphism analysis: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Dose Level 2: Patients receive temsirolimus IV over 30-60 minutes once weekly and bevacizumab IV over 30-90 minutes once every two weeks . Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  temsirolimus: Given IV
  bevacizumab: Given IV
  polymorphism analysis: Correlative studies
Arm/Group | Dose Level 1 | Dose Level 2
All-Cause Mortality (participants affected / at risk) | 1/4 | 7/20
Serious Adverse Events (participants affected / at risk) | 1/4 | 7/20
Other Adverse Events (participants affected / at risk) | 4/4 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=4) | Dose Level 2 (N=20)
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Pelvic (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Pain - Back (General disorders) | 0 (0) | 1 (1)
Pain - Extremity-limb (General disorders) | 0 (0) | 2 (2)
Pain - Pelvis (General disorders) | 0 (0) | 1 (1)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Weight loss (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=4) | Dose Level 2 (N=20)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 2 (4)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 2 (3)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 4 (4) | 12 (20)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 (0) | 4 (6)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (5) | 5 (16)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 2 (2) | 9 (12)
Conduction abnormality/atrioventricular heart block - Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (8)
Constitutional Symptoms - Cold intolerance (Psychiatric disorders) | 0 (0) | 1 (2)
Constitutional Symptoms - Change of mental sttatus (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 4 (6)
Dehydration (Gastrointestinal disorders) | 1 (1) | 3 (5)
Dental: periodontal disease (Gastrointestinal disorders) | 0 (0) | 3 (5)
Dermatology/Skin - hyperpigmentation-hands (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 5 (7)
Dizziness (Nervous system disorders) | 1 (1) | 4 (5)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Edema: limb (Vascular disorders) | 0 (0) | 7 (13)
Edema: trunk/genital (Vascular disorders) | 0 (0) | 1 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (10) | 12 (35)
Febrile neutropenia (ANC <1.0 x 10e9/L, fever >=38.5 degrees C) (Infections and infestations) | 1 (1) | 1 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 4 (4)
Fistula, GI - Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fistula, GI - Stomach (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal - early satiety (Gastrointestinal disorders) | 0 (0) | 1 (1)
rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1) | 8 (9)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 4 (14) | 9 (18)
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GU - Bladder (Renal and urinary disorders) | 0 (0) | 2 (3)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (11)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hot flashes/flushes (Endocrine disorders) | 0 (0) | 2 (3)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (2) | 3 (7)
Incontinence, anal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 0 (0) | 1 (2)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Insomnia (General disorders) | 0 (0) | 6 (6)
Joint-function (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (5) | 7 (16)
Lymphopenia (Blood and lymphatic system disorders) | 2 (12) | 15 (46)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 4 (8)
Mood alteration - Agitation (Nervous system disorders) | 0 (0) | 2 (3)
Mood alteration - Anxiety (Nervous system disorders) | 1 (1) | 2 (3)
Mood alteration - Depression (Nervous system disorders) | 1 (1) | 3 (4)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2 (5) | 5 (8)
Mucositis/stomatitis (functional/symptomatic) - Anus (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis/stomatitis (functional/symptomatic) - Esophagus (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 1 (1) | 8 (11)
Mucositis/stomatitis (functional/symptomatic) - Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extraocular (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscle weakness, generalized or specific area (not due to neuropathy) - Ocular (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Musculoskeletal/Soft Tissue -muscle aches in legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Nausea (Gastrointestinal disorders) | 3 (3) | 9 (19)
Neurology - decreased motivation (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 3 (6)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (4) | 3 (6)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 0 (0) | 2 (2)
Pain - Abdomen NOS (General disorders) | 0 (0) | 4 (5)
Pain - Anus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain - Back (General disorders) | 3 (5) | 6 (10)
Pain - Bone (General disorders) | 1 (1) | 2 (5)
Pain - Buttock (General disorders) | 0 (0) | 1 (1)
Pain - Chest wall (General disorders) | 2 (3) | 2 (2)
Pain - Chest/thorax NOS (General disorders) | 0 (0) | 1 (1)
Pain - Extremity-limb (General disorders) | 1 (1) | 6 (9)
Pain - Head/headache (General disorders) | 0 (0) | 3 (3)
Pain - Joint (General disorders) | 2 (2) | 8 (14)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (8)
Pain - Neck (General disorders) | 2 (5) | 1 (1)
Pain - Oral cavity (General disorders) | 0 (0) | 1 (2)
Pain - Diffuse pain;back,shoulders,hips,legs,ribs (General disorders) | 0 (0) | 1 (1)
Pain - L and R thigh (General disorders) | 0 (0) | 1 (1)
Pain - Pelvis (General disorders) | 1 (2) | 2 (3)
Pain - Peritoneum (General disorders) | 0 (0) | 1 (1)
Pain - Pleura (General disorders) | 0 (0) | 1 (1)
Pain - Throat/pharynx/larynx (General disorders) | 0 (0) | 3 (7)
Pain - Urethra (General disorders) | 0 (0) | 1 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Platelets (Blood and lymphatic system disorders) | 3 (6) | 10 (25)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) | 3 (9)
Proteinuria (Metabolism and nutrition disorders) | 2 (5) | 5 (5)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (7)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (7)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rigors/chills (General disorders) | 0 (0) | 2 (2)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) | 6 (9)
Sweating (diaphoresis) (General disorders) | 0 (0) | 2 (3)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (2) | 6 (13)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 3 (4) | 8 (12)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 8 (12)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 1 (1)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (7)
Watery eye (epiphora, tearing) (Eye disorders) | 0 (0) | 1 (1)
Weight loss (Gastrointestinal disorders) | 4 (4) | 9 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes